CLINICAL TRIAL: NCT02262299
Title: A European Multi-center, Randomised, Double-blind Trial of Pirfenidone in Bronchiolitis-obliterans-syndrome Grade 1-3 in Lung Transplant Recipients
Brief Title: European Trial of Pirfenidone in BOS, A European Multi-center Study
Acronym: EPOS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Perch, Medical Director Danish National Lung Transplant Program, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RH-HJE-2014-09
Record Dates: First submitted 2014-09-21; First posted 2014-10-13 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Disorder Related to Lung Transplantation; CLAD, Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Receive placebo tablets
  Interventions: Drug: Placebo
- Pirfenidone (Active Comparator): Upon enrollment, subjects will be randomized to either the treatment group (Pirfenidone) or to the placebo group (1:1 ratio). The trial medication will be administered as 267-mg oral capsules and titrated to a maintenance dose of 2403 mg/d (3 capsules TID, for a total of 9 capsules/day).
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Receive tablets with pirfenidone
  Other Names: Esbriet
  Arms: Pirfenidone
Drug: Placebo — Recieve tablets with placebo
  Arms: Placebo

SUMMARY:
A European multi-centre, randomised, double-blind placebo-controlled trial of Pirfenidone in bronchiolitis-obliterans-syndrome grade 1-3 in lung transplant recipients.

Randomized double blinded, placebo controlled study. Eligible patients are to be randomized in a 1:1 ratio to receive either Pirfenidone 2403 mg/d or the matching placebo treatment for 6 months.

Primary objective To evaluate the effect of Pirfenidone on the change in FEV1 in liters over 6 months in lung transplant recipients with bronchiolitis obliterans syndrome.

DETAILED DESCRIPTION:
Title of the study: A European multi-centre, randomised, double-blind placebo-controlled trial of Pirfenidone in bronchiolitis-obliterans-syndrome grade 1-3 in lung transplant recipients

Study design: Randomized double blinded, placebo controlled study. Eligible patients are to be randomized in a 1:1 ratio to receive either Pirfenidone 2403 mg/d or the matching placebo treatment for 6 months.

Study objectives Primary objective:

Change in FEV1 in liters over 6 months in lung transplant recipients with bronchiolitis obliterans syndrome.

Secondary objectives:

* Categorical percentage change in FEV1
* Change in Forced Vital Capacity (FVC)
* Change in Total Lung Capacity (TLC)
* Change in FEV1/FVC ratio
* Number of patients with treatment failure
* Change in BOS grade
* Change in percent predicted diffusion capacity (DLCO)
* Change in functional level as assessed by the 6MWT
* Hospital admission for any reason
* Death or re-transplantation rates
* Change in QoL as assessed by EQ5D

Methodology The study will be conducted in selected Lung Transplant expert centers across Europe.

Trial duration Enrolment duration: planned 15 months Treatment duration: 6 months

Number of patients Number of sites Number of countries ~80 patients ( ~40 per Arm) A minimum of 10 centers 7 (Denmark, Sweden, Norway, UK, Belgium, The Netherlands and Germany)

Study treatment: Patients will be randomized 1:1 to receive either placebo or Pirfenidone.

Pirfenidone dose will be adapted per the Investigator's Brochure in case of adverse events

Selection criteria: Inclusion criteria:

Patients can be included irrespective of pre-transplant disease, type of induction treatment and immunosuppressive treatment. The following patients will be included in the study:

* Patients >18 years of age
* Azithromycin therapy for at least 4 weeks prior to study start, with an Azithromycin dose of minimum 250 mg/day at least 3 times per week as this is considered standard therapy for bronchiolitis obliterans syndrome.
* Double lung transplantation is required.
* Patients must be at least 6 months after transplantation and must have documented post-transplant baseline value of FEV1 (mean of the 2 highest values measured at least 3 weeks apart according to ISHLT criteria).
* Patients must have BOS grade 1 to BOS grade 3.
* Patients must have documented progressive disease as demonstrated by all of the following criteria:
* Patients must have at least 3 FEV1-measurements in the last 6 months, each at least 3 weeks apart
* a total decline of at least 200ml in FEV1 in these last three measurements
* a decline of at least 50 ml in the last two measurements

Exclusion Criteria:

* Patients with lung redo transplantation, combined transplantation (including heart and lung transplantation) or single lung recipients.
* Patients with any severe comorbidity complicating BOS which might determine the prognosis and functional level of the patient (e.g. invasive aspergillosis, active malignant disease) within the last 12 months.
* FEV1 decline related to other non BOS causes (eg pneumothorax, bronchial stenosis, effusion, etc.)
* Patients who on Thorax CT at entry demonstrate new significant findings which are not compatible with BOS like interstitial fibrosis, consolidation, appearances suggesting Restrictive Allograft Syndrome (RAS) and acute pulmonary infection as cause of decline in lung function.
* Documented acute perivascular rejection higher than grade A1 or findings compatible with antibody mediated rejection
* Pregnancy or lactation (women of childbearing capacity are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of the study).
* Renal insufficiency (Creatinine clearance <30 ml/min calculated by the CKD-Epi formula.
* Any of the following liver test criteria above the specified limit:
* Total bilirubin above the upper limit of the normal range (ULN), except in patients with predominantly unconjugated hyperbilirubinemia (e.g., Gilbert's syndrome)
* Aspartate or alanine aminotransferase (AST or ALT) >3 × ULN
* Known allergy or hypersensitivity to Pirfenidone
* Ongoing use or expected use of any of the following therapies:
* Strong inhibitors of CYP1A2 (e.g. fluvoxamine or enoxacin)
* Moderate inhibitors of CYP1A2 (e.g. mexiletine, thiabendazole, or phenylpropanolamine [Note: ciprofloxacin will be allowed only at doses ≤500 mg BID])
* Previous treatment with Pirfenidone after transplantation
* Patients who have resumed smoking after transplantation

Data collection At screening:

* Thorax HR-CT ( to exclude non-BOS pathology)
* Chest X Ray
* Spirometry and measurement of FEV1/FVC according to ERS criteria is required to demonstrate typical obstruction
* ECG to exclude QTc > 500ms
* Bronchoscopy with bronchoalveolar lavage (BAL) according to standard international criteria. At least two aliquots of 50 ml are required. BAL to exclude concurrent infections. BAL cultured for bacteria and fungi plus cytospin preparations or immunological BAL for differential counts.
* Transbronchial biopsy
* Blood samples (haematology and chemistry) including liver function tests
* Drug monitoring for immuno-suppressive treatment

Baseline:

* Height
* Weight
* Basic demographic data including medication.
* Physical examination and vital signs
* Spirometry and measurement of FEV1/FVC
* Blood samples (haematology and chemistry) including liver function tests
* Drug monitoring for immuno-suppressive treatment
* Record concomitant medications
* Body-plethysmographic measurement to assess TLC and RV
* DLco
* 6MWT
* Quality of Life questionnaire

Monthly visits (Months 1, 2, 3, 4):

* Weight
* Spirometry and measurement of FEV1/FVC according to ATS/ERS criteria.
* Safety monitoring (Record ADRs and blood lab tests, including liver tests)
* Drug monitoring for immuno-suppressive treatment
* Record concomitant medications
* Clinical Status

Endpoints: 6 Month visit (or early termination visit):

* Weight
* Spirometry and measurement of FEV1/FVC according to ATS/ERS criteria.
* Safety monitoring (Record ADRs and blood lab tests, including liver tests)
* Drug monitoring for immuno-suppressive treatment
* Record concomitant medications
* Clinical Status
* Body-plethysmographic measurement to assess TLC and RV
* DLco
* 6MWT
* Quality of Life questionnaire

Primary endpoints

- Change in FEV1 (ml) at 6 months

Secondary endpoints

* Categorical percentage change in FEV1 (ml)

  o Categorical percentage change in FEV1 ≥ 10 % (increase or decrease) relative to FEV1(ml) at baseline
* Change of FVC in liters
* Change in TLC in liters
* FEV1/FVC ratio change
* Number of patients with treatment failure
* Change in BOS grade
* Change in percent predicted DLco.
* Change in functional level as assessed by the 6MWT
* Hospital admission for any reason
* Death or re-transplantation rates
* Change in EQ5D scale

Treatment failure during the study is defined as one or more of the following:

* Redo transplantation
* Death due to respiratory causes
* Initiation of rescue therapy for worsening of BOS (worsening of BOS defined as a decline of at least 600mL in 3 consecutive months) o Photophoresis, Montelukast or other treatment considered as rescue therapy by the investigator

Statistical Methods Imputation:

In the ITT primary endpoint analysis, missing data due to treatment failure and death will be imputed as 50% of baseline FEV1. For patients lost to follow-up or who withdrew from the study for reasons not related to BOS, the last measured FEV1 (ml) will be imputed as the 6 month value.

Sample Size calculation:

Assumptions:

1. SD: To determine the SD of the FEV1 decline in the population, the 5 members of the Steering committee collected the data from patients meeting the inclusion criteria. Mean decline in FEV1 (in a 6 month period) in this sample was 561 ml and the SD of the decline was 300 ml .
2. Treatment effect: A meaningful treatment effect of 50% should be expected based on the mechanism of disease and preliminary data in BOS (In the publication) and personal experience.

One standard deviation (SD) of FEV1 in groups will be assumed to be 300 mL based on data from expert centers.

Monthly decline in FEV1 at onset of BOS is assumed to be approximately 75 ml, in 6 months 450 ml decline in FEV1 is expected for the placebo group.

A treatment effect of 50% reduction in decline is expected with Pirfenidone, which will lead to an expected mean decline of 225 ml in 6 months.

With a beta error of 12% (power 88%) the study will be able to detect a difference of 225 ml between the two treatment groups with a sample size of 36 patients in each group using a two-sided t-test with significance level of 0.05. An estimated 80 patients will be recruited to the trial allowing for a drop-out rate of 10%.

Concomitant treatment - Stopping Azithromycin will be allowed if not tolerated. Standard treatment is continuation of Azithromycin.

* Initiation on new bronchodilator therapy is not allowed
* Photopheresis and Montelukast are not allowed while on Pirfenidone Study Committees Steering Committee: M. Perch, P. Corris, G. Verleden, J. Gotlieb and E Verschuuren Patient Review Committee Inclusion Criteria, exclusion criteria and BOS staging for all patients enrolled will be reviewed by a committee.

Clinical Events Committee Group of physicians who will review the serious adverse events that occur during the study to adjudicate their relationship to the study drug.

DSMB Independent group to review the safety and efficacy data during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Azithromycin therapy for at least 4 weeks prior to study start, with an Azithromycin dose of minimum 250 mg/day at least 3 times per week as this is considered standard therapy for bronchiolitis obliterans syndrome.
* Double lung transplantation is required.
* Patients must be at least 6 months after transplantation and must have documented post-transplant baseline value of FEV1 (mean of the 2 highest values measured at least 3 weeks apart according to ISHLT criteria).
* Patients must have BOS grade 1 to BOS grade 3.
* Patients must have documented progressive disease as demonstrated by all of the following criteria:
* Patients must have at least 3 FEV1-measurements in the last 6 months, each at least 3 weeks apart
* a total decline of at least 200ml in FEV1 i
* a decline of at least 50 ml in the last two measurements

Exclusion Criteria

* Patients with lung redo transplantation, combined transplantation (including heart and lung transplantation) or single lung recipients.
* Patients with any severe comorbidity complicating BOS which might determine the prognosis and functional level of the patient (e.g. invasive aspergillosis, active malignant disease) within the last 12 months.
* FEV1 decline related to other non BOS causes (eg pneumothorax, bronchial stenosis, effusion, etc.)
* Patients who have developed BOS grade 3.
* Patients who on Thorax CT at entry demonstrate new significant findings which are not compatible with BOS like interstitial fibrosis, consolidation, appearances suggesting Restrictive Allograft Syndrome (RAS) and acute pulmonary infection as cause of decline in lung function.
* Documented acute perivascular rejection higher than grade A1 or findings compatible with antibody mediated rejection
* Pregnancy or lactation (women of childbearing capacity are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using at least two methods of birth control from the date of consent through the end of the study).
* Renal insufficiency (Creatinine clearance <30 ml/min calculated by the CKD-Epi formula.
* Any of the following liver test criteria above the specified limit:
* Total bilirubin above the upper limit of the normal range (ULN), except in patients with predominantly unconjugated hyperbilirubinemia (e.g., Gilbert's syndrome)
* Aspartate or alanine aminotransferase (AST or ALT) >3 × ULN
* Known allergy or hypersensitivity to Pirfenidone
* Ongoing use or expected use of any of the following therapies:
* Strong inhibitors of CYP1A2 (e.g. fluvoxamine or enoxacin)
* Moderate inhibitors of CYP1A2 (e.g. mexiletine, thiabendazole, or phenylpropanolamine [Note: ciprofloxacin will be allowed only at doses ≤500 mg BID])
* Previous treatment with Pirfenidone after transplantation
* Patients who have resumed smoking after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Pirfenidone on the change in FEV1 in liters over 6 months in lung transplant recipients with bronchiolitis obliterans syndrome. | 6 months

SECONDARY OUTCOMES:
- Categorical percentage change in FEV1 | 6 months
- Change in Forced Vital Capacity (FVC) | 6 months
- Change in Total Lung Capacity (TLC) | 6 months
- Change in FEV1/FVC ratio | 6 months
- Number of patients with treatment failure | 6 months
- Change in BOS grade | 6 months
- Change in percent predicted diffusion capacity (DLCO) | 6 months
- Change in functional level as assessed by the 6MWT | 6 months
- Hospital admission for any reason | 6 months
- Death or re-transplantation rates | 6 months
- Change in QoL as assessed by EQ5D | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perch, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (9):
- University Hospital Gasthuisberg, Katholike Universiteit Leuven, Leuven, Belgium
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- Germany (3):
  - University Hospital Essen, Department of Pneumonology, Essen
  - Medizinische Hochschule Hannover, Klinik für Pneumonologie, Hanover
  - Klinikum Grosshadern, Division of Pulmonary Diseases, Munich
- Groningen University Medical Center, Lung Transplant Team, Groningen, Netherlands
- Rikshospitalet, National University Hospital, Oslo, Norway
- Sahlgrenska University Hospital, Department of respiratory diseases, Gothenburg, Sweden
- Freeman Hospital, Newcastle, United Kingdom

REFERENCES:
- [Derived] Perch M, Corris P, Lordan J, Bessa V, Magnusson J, Verleden GM, Vos R, Kneidinger N, Leuckfeld I, Verschuuren E, Gottlieb J. A European multi-center, randomized controlled trial of Pirfenidone in bronchiolitis obliterans syndrome after bilateral lung transplantation. Eur Respir J. 2025 Nov 13:2402154. doi: 10.1183/13993003.02154-2024. Online ahead of print. PMID 41232942